CLINICAL TRIAL: NCT06086080
Title: Non-operative Treatment in First-time Patellar Dislocation: a Randomized Controlled Trial
Brief Title: Non-operative Treatment in First-time Patellar Dislocation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinica Valle del Lili (Other)
Collaborators: International Society of Arthroscopy, Knee Surgery and Orthopaedic Sports Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 1906
Record Dates: First submitted 2023-10-03; First posted 2023-10-17 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Patellar Dislocation
Keywords: Patellar dislocation; Brace; Knee taping
MeSH Terms: conditions — Patellar Dislocation | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients are randomized either to standard care or in the intervention group. Standard care patients are treated with knee brace (2 weeks) and physical therapy. In the intervention group: they receive knee taping with knee brace during 1-week.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcomes assessor will not have access to the type of treatment a patient received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Standard care: knee brace for 2 weeks, physical therapy, sham taping (2-weeks)
  Interventions: Other: Standard care; Device: Sham taping
- Intervention group (Experimental): Knee taping for 4-weeks, knee brace for 1 week, physical therapy
  Interventions: Other: Standard care; Other: Taping

INTERVENTIONS:
Other: Standard care — Bracing and physical therapy
Other: Taping — The patient is treated with tape in special configuration (McConell modified) for the patella + standard care
  Arms: Intervention group
Device: Sham taping — Taping with no treatment disposition
  Arms: Control group

SUMMARY:
Study to evaluate the conservative treatment of patients after their first episode of primary lateral patellar dislocation. Randomized controlled trial with 2 groups: standard treatment (2-weeks with brace) followed by physical therapy, compared with knee taping and physical therapy. 1-year follow-up. Measurements include physical exam, radiographs and MRI. Outcomes: recurrence, lateral patellar tilt, functional scores, apprehension, pain.

Hypothesis: less recurrence in the knee taping group, as well as better functional scores.

DETAILED DESCRIPTION:
Patients between 10-40 years old with first patellar dislocation are invited to participate in this conservative treatment study.

Patients are excluded if they have bilateral acute patellar dislocation, previous surgeries in the affected knee, osteochondral fracture, open patellar dislocation.

This is a randomized controlled trial with four groups of treatment:

1. Standard treatment (2-weeks with a knee brace) and physical therapy
2. Knee taping and physical therapy (1-week with knee brace)

Sample size: 50 patients / knees Outcomes of interest: recurrence in patellar dislocation, functional scores (Banff, Norwich), return to sport, patellar tilt

ELIGIBILITY:
Inclusion Criteria:

- Patients with first episode of acute lateral patellar dislocation during the last 7 days.

Exclusion Criteria:

* Patients with acute bilateral patellar dislocation.

* Patients with open patellar dislocation.
* Patients with previous knee surgery in the same knee.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Recurrent patellar dislocation (percentage of patients) | 2 years
  Percentage of patients with additional patellar dislocation after the first episode

SECONDARY OUTCOMES:
Banff Patellofemoral Instability Instrument (BPII) | 2 years
  Patellofemoral instability specific score to assess function (disease-specific). The punctuation range is between 0-100 points. The best health scenario is 100% and the worst is 0.
Nich patellar instability (NPI) score | 2 years
  Patellofemoral instability specific score to assess function (disease-specific). The punctuation range is between 0-100%. The worst health deficit is 100% and the best is 0%.

OTHER OUTCOMES:
Patellar tilt angle of patients after the first episode | 1 month
  Patellar tilt in magnetic resonance imaging (angle in degrees)
Patellar apprehension test | 2 years
  Patellar apprehension test during physical examination. The quadriceps should be relaxed to allow passive movements of the patella. The clinician will perform this technique by using their thumb of both hands, and pressing on the medial side of the patient's patella. The test is positive if it produces pain and apprehension.
Percentage of participants with patellar J sign | 2 years
  J sign during physical examination. The J-sign refers to the inverted 'J' track the patella takes from extension to early flexion. The J-sign is a clinical finding indicative of patellar maltracking.
Percentage of participants that return to sport activity | 2 years
  Percentage of the patients that were able to return to do their usual sport after the initial injury (patellar dislocation)

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Martinez, MD, Principal Investigator — Fundacion Clinica Valle del Lili
Locations (1):
- Fundación Valle del Lili, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: For 5 years after publishing the paper.
Access Criteria: Data will be shared if it is found to be relevant for understanding better the study or the analysis. This includes the journal where the paper is submitted and investigators with interest in the study.